CLINICAL TRIAL: NCT04132219
Title: Daughters, (dUdes), Mothers and othErs Fighting Cancer Together
Brief Title: Daughters, dUdes, Mothers and othErs Fighting Cancer Together
Acronym: DUET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Wendy Demark-Wahnefried, PhD, Professor and Webb Endowed Chair of Nutrition Sciences, University of Alabama at Birmingham (UAB) Associate Director of Cancer Prevention and Control, O'Neal Comprehensive Cancer Center, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-300003882
Record Dates: First submitted 2019-10-11; First posted 2019-10-18 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-05

CONDITIONS: Cancer; Overweight and Obesity
Keywords: cancer survivor; overweight; obesity
MeSH Terms: conditions — Neoplasms; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: We anticipate enrolling 56 dyads of participants (2 per dyad). Each dyad will be randomized to either receive the intervention for 6 months or be placed on a 6-month waitlist and offered the opportunity to try the online intervention after final assessments are completed.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors of anthropometric, physical function, patient reported outcomes and biospecimens are blinded to arm status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Dyads randomized to the Immediate Intervention Group will receive a "Welcome Box" at completion of the baseline assessment. The Welcome Box will include two of each of the following: 1) Letters describing the project logistics and the important roles of each dyad member); 2) WiFi-enabled Scales (with instructions to weigh daily); 3) Portion Doctor ®Tableware (with instructions to use the portion plates at least once a day); 4) Fitbit® Inspire Activity Monitors (with instructions to share data with the dyad member and the study office); and 5) Instructions on how to create a secured account on the DUET website and instructions for logging on.
  Interventions: Behavioral: eHealth Intervention
- Delayed Intervention Group (Other): Participants assigned to the Delayed Intervention Group will receive a "Welcome Box" which on the outside is identical (and also is comparably weighted with bottled water) to that given to the Immediate Intervention group. This box would include: 1) Letters describing the project logistics and the important roles of each dyad member; and 2) monthly online study newsletters on topics unrelated to diet and exercise, but still of interest to cancer survivors and dyad members such as coping with stress, reducing exposure to radiation, sun safety, etc. to enhance retention and will be offered the opportunity to receive the online intervention after completing final 6-month assessments.
  Interventions: Behavioral: eHealth Intervention

INTERVENTIONS:
Behavioral: eHealth Intervention — Every week, each dyad member will receive a tailored text message that provides a new fun fact or that encourages them to log-on to the website to access findings of new research and how the results might apply to them. They will be directed to specific pages in the Web-based program and asked to select strategies from a list that they will practice during the upcoming week. Graphic displays of their progress will be provided along with SCT-based feedback. They will be directed to the website to record their behavioral goals for the upcoming week. Tips also will be provided for effective communication to enhance couple efficacy. All usage will be tracked to assess adherence.

SUMMARY:
The purpose of this protocol is to conduct a 2-arm, single-blinded randomized controlled clinical trial (RCT) in which 56 dyads (defined as consisting of an overweight or obese cancer survivor of an obesity-related cancer and an overweight or obese "buddy" of his or her choosing) would be assigned either to a 6-month, diet- and exercise-based weight loss intervention delivered via an interactive website with tailored text messages, or to a 6-month wait-listed control group. The overall goals of the eHealth intervention are to reduce obesity and select circulating biomarkers (tumor necrosis factor alpha [TNFα], insulin, and insulin-like growth factor-1 [IGF-1]), as well as improve diet quality, physical activity, health-related quality of life (QoL), physical functioning and performance as compared to the control over the 6-month study period.

DETAILED DESCRIPTION:
The specific aims of this protocol are to: 1) determine whether dyads (comprised of an overweight / obese cancer survivor and an overweight / obese buddy of his or her choosing) lose significantly more weight (kg) at 6-months when assigned to the eHealth intervention compared to a wait-listed control; 2) explore between-arm differences in score changes between baseline and 6-month follow-up for other key outcomes including measures of adiposity (e.g., waist circumference [WC] and body mass index [BMI]), blood pressure, diet quality, physical activity, health-related Quality of Life (QoL), physical functioning and performance; 3) Assess the impact of the intervention on select biomarkers associated with cancer risk and progression, e.g., tumor TNFα, insulin and IGF-1; and, 4) identify predictor variables associated with program efficacy, e.g., social support, self-efficacy, risk for depression, and dyad partner (spouse, relative, friend/neighbor).

Cancer survivors and their selected "buddies" who are interested in participating will be directed to a website that describes this study in detail. If interested, they will be asked to complete an online screener requiring information on race/ethnicity, gender, state of residence and eligibility criteria. Once interested participants are assessed for eligibility, consented and enrolled, they will be asked to complete online questionnaires that assess physical activity, dietary intake, health-related quality of life, risk for depression, self-efficacy, social support and barriers to diet resources. Finally, anthropometric measures, blood pressure, physical performance and circulating biomarkers will be collected in participants' homes by visiting study staff (whom the project manager will deploy after checking for a mutually convenient time for the 2-person dyad.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18+ for whom at least one dyad member has been diagnosed and completed curative treatment for localized renal cancer, or loco-regional ovarian, colorectal, endometrial, or female breast cancer. (Loco-regional prostate cancer survivors are also eligible but could be on active surveillance).
* Diagnosed as overweight or obese (BMI >25 kg/m2.
* Low vegetable and fruit intake (<2.5 cups day).
* Low physical activity (<150 minutes per week).
* English-speaking and writing.
* Completed at least 5th grade.
* Uses the internet and owns a mobile phone.

Exclusion Criteria:

* Diagnosed with uncontrolled chronic conditions (i.e., diabetes, blood pressure, CVD, etc)
* Diagnosed with a health conditions that precludes adherence to an unsupervised weight loss intervention (e.g., pregnancy, end-stage renal disease, etc).
* Instructed by a physician to limit physical activity AND have paralysis, dementia, blindness, unstable angina, untreated stage 3 hypertension, or recent history of heart attack, congestive heart failure or pulmonary conditions that required oxygen or hospitalization within 6 months.
* Diagnosed with other cancers (except non-malignant skin cancer), cancer recurrence or metastatic disease.
* Resides in a skilled nursing or assisted living facility.
* Resides more than 15 minute driving distance from dyad partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Body Weight | baseline
  Change in measured body weight
Body Weight | 6 months
  Change in measured body weight

SECONDARY OUTCOMES:
Waist Circumference | baseline
  measured with a non-stretch tape
Waist Circumference | 6 months
  measured with a non-stretch tape
Physical Activity (self-reported) | Baseline
  Godin Leisure Time Physical Activity Questionnaire (4-item survey) - individuals provide the number of minutes of vigorous, moderate and light physical activity per week. The minimum is 0 - theoretically, the maximum is 10,080 (the number of minutes in a week), then they are asked if this level of activity is "typical." The higher the number of minutes of totaled moderate + vigorous activity, the better.
Physical Activity (self-reported) | 3 months
  Godin Leisure Time Physical Activity Questionnaire (4-item survey) - individuals provide the number of minutes of vigorous, moderate and light physical activity per week. The minimum is 0 - theoretically, the maximum is 10,080 (the number of minutes in a week), then they are asked if this level of activity is "typical." The higher the number of minutes of totaled moderate + vigorous activity, the better.
Physical Activity (self-reported) | 6 months
  Godin Leisure Time Physical Activity Questionnaire (4-item survey) - individuals provide the number of minutes of vigorous, moderate and light physical activity per week. The minimum is 0 - theoretically, the maximum is 10,080 (the number of minutes in a week), then they are asked if this level of activity is "typical." The higher the number of minutes of totaled moderate + vigorous activity, the better.
Physical Activity (objective) | baseline
  Accelerometry (7-day assessment)
Physical Activity (objective) | 6 months
  Accelerometry (7-day assessment)
Diet Quality | baseline
  Two 24-hour dietary recalls
Diet Quality | 6 months
  Two 24-hour dietary recalls
Physical Performance (endurance) | Baseline
  2-minute step test
Physical Performance (endurance) | 6 months
  2-minute step test
Physical Performance (lower body strength) | Baseline
  30-second chair stand
Physical Performance (lower body strength) | 6 months
  30-second chair stand
Physical Performance (agility) | Baseline
  8' foot up and go
Physical Performance (agility) | 6 months
  8' foot up and go
Physical Performance (gait speed) | baseline
  8' walk
Physical Performance (gait speed) | 6 months
  8' walk
Physical Performance (Balance) | baseline
  Side-by-side, semi-tandem and tandem stances
Physical Performance (Balance) | 6 months
  Side-by-side, semi-tandem and tandem stances
Self-efficacy for calorically restricted diet | baseline
  Clark et al. survey (20 items). Respondents either affirm or deny that they can resist high fat, high calorie foods under a variety of situations. Individuals who have maximum willpower achieve the top score of 20, whereas those with lesser willpower score lower (the minimum score is zero)
Self-efficacy for calorically restricted diet | 3 months
  Clark et al. survey (20 items). Respondents either affirm or deny that they can resist high fat, high calorie foods under a variety of situations. Individuals who have maximum willpower achieve the top score of 20, whereas those with lesser willpower score lower (the minimum score is zero)
Self-efficacy for calorically restricted diet | 6 months
  Clark et al. survey (20 items). Respondents either affirm or deny that they can resist high fat, high calorie foods under a variety of situations. Individuals who have maximum willpower achieve the top score of 20, whereas those with lesser willpower score lower (the minimum score is zero)
Self-efficacy for increased physical activity | baseline
  Sallis et al. survey (6 items in total). Respondents rate themselves on each item from 0 to 100% on their level of confidence. The higher the total score (maximum of 100%) the better (Minimum 0%).
Self-efficacy for increased physical activity | 3 months
  Sallis et al. survey (6 items in total). Respondents rate themselves on each item from 0 to 100% on their level of confidence. The higher the total score (maximum of 100%) the better (Minimum 0%).
Self-efficacy for increased physical activity | 6 months
  Sallis et al. survey (6 items in total). Respondents rate themselves on each item from 0 to 100% on their level of confidence. The higher the total score (maximum of 100%) the better (Minimum 0%).
Social support for calorically restricted diet | baseline
  Sallis et al. instrument (4 items). Respondents rate the level of support they obtain to follow a healthy, low calorie diet on a 5-point scale ranging from ("never"= 0 to "everyday" = 4. Individuals who have maximum support achieve the top score of 16, whereas those with lesser support score lower (the minimum score is zero)
Social support for increased physical activity | baseline
  Sallis et al. instrument (4 items in total) Respondents rate the level of support they obtain to increase their level of physical activity on a 5-point scale ranging from ("never"= 0 to "everyday" = 4. Individuals who have maximum support achieve the top score of 16, whereas those with lesser support score lower (the minimum score is zero)
Social support for calorically restricted diet | 3 months
  Sallis et al. instrument (4 items). Respondents rate the level of support they obtain to follow a healthy, low calorie diet on a 5-point scale ranging from ("never"= 0 to "everyday" = 4. Individuals who have maximum support achieve the top score of 16, whereas those with lesser support score lower (the minimum score is zero)
Social support for increased physical activity | 3 months
  Sallis et al. instrument (4 items in total) Respondents rate the level of support they obtain to increase their level of physical activity on a 5-point scale ranging from ("never"= 0 to "everyday" = 4. Individuals who have maximum support achieve the top score of 16, whereas those with lesser support score lower (the minimum score is zero)
Social support for calorically restricted diet | 6 months
  Sallis et al. instrument (4 items). Respondents rate the level of support they obtain to follow a healthy, low calorie diet on a 5-point scale ranging from ("never"= 0 to "everyday" = 4. Individuals who have maximum support achieve the top score of 16, whereas those with lesser support score lower (the minimum score is zero)
Social support for increased physical activity | 6 months
  Sallis et al. instrument (4 items in total) Respondents rate the level of support they obtain to increase their level of physical activity on a 5-point scale ranging from ("never"= 0 to "everyday" = 4. Individuals who have maximum support achieve the top score of 16, whereas those with lesser support score lower (the minimum score is zero)
Barriers for increased physical activity | baseline
  (15 items in total) Respondents either affirm or deny common barriers to exercise. Individuals who report more barriers achieve the top score of 21, whereas those with fewer barriers score lower (the minimum score is zero) and that is considered better.
Barriers for increased physical activity | 3 months
  (15 items in total) Respondents either affirm or deny common barriers to exercise. Individuals who report more barriers achieve the top score of 21, whereas those with fewer barriers score lower (the minimum score is zero) and that is considered better.
Barriers for increased physical activity | 6 months
  (15 items in total) Respondents either affirm or deny common barriers to exercise. Individuals who report more barriers achieve the top score of 21, whereas those with fewer barriers score lower (the minimum score is zero) and that is considered better.
Circulating insulin | baseline
  assays on dried blood spot eluents
Circulating insulin | 6 months
  assays on dried blood spot eluents
Circulating glucose | baseline
  assays on dried blood spot eluents
Circulating glucose | 6 months
  assays on dried blood spot eluents
Circulating IL-6 | baseline
  assays on dried blood spot eluents
Circulating IL-6 | 6 months
  assays on dried blood spot eluents
Circulating CRP | baseline
  assays on dried blood spot eluents
Circulating CRP | 6 months
  assays on dried blood spot eluents
Circulating Total Cholesterol | baseline
  assays on dried blood spot eluents
Circulating Total Cholesterol | 6 months
  assays on dried blood spot eluents
Circulating HDL Cholesterol | baseline
  assays on dried blood spot eluents
Circulating HDL Cholesterol | 6 months
  assays on dried blood spot eluents
Circulating Tryglycerides | baseline
  assays on dried blood spot eluents
Circulating Tryglycerides | 6 months
  assays on dried blood spot eluents
Circulating Adiponectin | baseline
  assays on dried blood spot eluents
Circulating Adiponectin | 6 months
  assays on dried blood spot eluents
Circulating Leptin | baseline
  assays on dried blood spot eluents
Circulating Leptin | 6 months
  assays on dried blood spot eluents
Duke OARS Co-Morbidity Index | baseline
  43-item assessment of co-morbid conditions (multiple choice) (modified by removing 1 item)
Duke OARS Co-Morbidity Index | 3 months
  43-item assessment of co-morbid conditions (multiple choice) (modified by removing 1 item)
Duke OARS Co-Morbidity Index | 6 months
  43-item assessment of co-morbid conditions (multiple choice) (modified by removing 1 item)
PROMIS v.1.2 GLOBAL HEALTH | Baseline
  10-item Likert scale assessment of Quality of Life
PROMIS v.1.2 GLOBAL HEALTH | 3 months
  10-item Likert scale assessment of Quality of Life
PROMIS v.1.2 GLOBAL HEALTH | 6 months
  10-item Likert scale assessment of Quality of Life
EQ-5D-5L | Baseline
  6-item Likert scale assessment of Quality of Life
EQ-5D-5L | 3 months
  6-item Likert scale assessment of Quality of Life
EQ-5D-5L | 6 months
  6-item Likert scale assessment of Quality of Life
HEALTH / E-HEALTH LITERACY SCALE (NORMAN 2006) | Baseline
  7-item scale to assess e-health literacy. Two items were added from eHEALS to understand consumer's interest in using eHealth in general.
HEALTH / E-HEALTH LITERACY SCALE (NORMAN 2006) | 3 months
  7-item scale to assess health and e-health literacy. Two items were added from eHEALS to understand consumer's interest in using eHealth in general.
HEALTH / E-HEALTH LITERACY SCALE (NORMAN 2006) | 6 months
  7-item scale to assess health and e-health literacy. Two items were added from eHEALS to understand consumer's interest in using eHealth in general.
Barriers to Eating a Healthy Low Calorie Diet | Baseline
  (10 items) Respondents either affirm or deny common barriers to low calorie diet.
Barriers to Eating a Healthy Low Calorie Diet | 3 months
  (10 items) Respondents either affirm or deny common barriers to low calorie diet.
Barriers to Eating a Healthy Low Calorie Diet | 6 months
  (10 items) Respondents either affirm or deny common barriers to low calorie diet.
PROMIS Emotional Distress: Depression - Short Form 8a | Baseline
  (8 items) Likert scale assessment of depression
PROMIS Emotional Distress: Depression - Short Form 8a | 3 months
  (8 items) Likert scale assessment of depression
PROMIS Emotional Distress: Depression - Short Form 8a | 6 months
  (8 items) Likert scale assessment of depression
Smoking status | Baseline
  2 items that ask whether respondent has ever smoked >100 cigarettes and current smoking status.
Smoking status | 3 months
  2 items that ask whether respondent has ever smoked >100 cigarettes and current smoking status.
Smoking status | 6 months
  2 items that ask whether respondent has ever smoked >100 cigarettes and current smoking status.

OTHER OUTCOMES:
Relationship to chosen partner | Baseline
  1 item question that asks for relationship of chosen partner to cancer survivor
Socio-Demographic (George, et al, 1984) | Baseline
  3-items that ask about income and perceptions of economic well-being
Socio-Demographic (George, et al, 1984) | 3 months
  3-items that ask about income and perceptions of economic well-being
Socio-Demographic (George, et al, 1984) | 6 months
  3-items that ask about income and perceptions of economic well-being
Circulating Insulin (TSH) | Baseline
  assays on dried blood spot eluents
Circulating Insulin (TSH) | 6 months
  assays on dried blood spot eluents

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, RD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB School of Health Professions, Department of Nutrition Sciences, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at the moment to share IDP.

REFERENCES:
- [Background] Pekmezi DW, Crane TE, Oster RA, Rogers LQ, Hoenemeyer T, Farrell D, Cole WW, Wolin K, Badr H, Demark-Wahnefried W. Rationale and Methods for a Randomized Controlled Trial of a Dyadic, Web-Based, Weight Loss Intervention among Cancer Survivors and Partners: The DUET Study. Nutrients. 2021 Sep 29;13(10):3472. doi: 10.3390/nu13103472. PMID 34684474
- [Derived] Kaur H, Pekmezi D, E Crane T, Farrell D, Q Rogers L, Demark-Wahnefried W. Website Use and Associations With Behavior Change and Weight Loss in Cancer Survivors and Their Partners: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2026 Jan 30;28:e86908. doi: 10.2196/86908. PMID 41617212
- [Derived] Kaur H, Pavela G, Pekmezi DW, Rogers LQ, Cole WW, Parrish KB, Sayer RD, Wyatt HR, Crane TE, Badr H, Demark-Wahnefried W. Living together-does it help or hinder the pursuit of a healthful diet, physical activity, and weight loss among cancer survivors and their chosen partners? Support Care Cancer. 2024 Oct 3;32(10):700. doi: 10.1007/s00520-024-08907-3. PMID 39361227